CLINICAL TRIAL: NCT03353805
Title: Hospital Cohort Survey of Public Health Post-attack of July 14, 2016
Acronym: ECHOS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 17-PP-05
Record Dates: First submitted 2017-11-17; First posted 2017-11-27 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Mental Disorders; Psychological Trauma
MeSH Terms: conditions — Mental Disorders; Psychological Trauma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaire — questionnaire

SUMMARY:
The terrorist attack on the ram truck, which occurred on 14 July 2016 on the Promenade des Anglais in Nice, involved a significant number of casualties in the civilian population: 86 dead including 10 children and adolescents, and 434 wounded. The attack harmed families gathered for a festive event, the national holiday fireworks, and affected both adults and children of all ages. The people directly involved in the attack number in the thousands: wounded, threatened with death, bereaved, direct witnesses, workers - including firefighters and health personnel (in situations of prolonged extreme tension or insecurity).

Following the attacks in Ile-de-France in January and November 2015, Public Health France conducted in 2015 and 2016 two large-scale studies to estimate the psycho-traumatic impact for those involved in the attack, to know the use of care devices to provide useful information, and ultimately provide information to improve the management devices in place. IMPACTS carried out following the attacks of January, ESPA 13 November carried out following the attacks of 13 November 2015, relate to two main types of population:

* Non-responders (civilian population) present on or near scenes of crime or their relatives.
* Persons intervened to secure the premises or provide assistance, or provide psychological support the same day or within 3 weeks.

IMPACTS was conducted face-to-face with investigators and concerned 232 participants, 45 people of the medico-psychological relief (Samu, Cump, Hôtel Dieu) between 6 and 10 months after the events. A second wave of interviews took place from 16 to 20 months after the events.

ESPA 13th November took place via a web-based questionnaire and 800 participants took part, including 67 CUMPs, 121 hospital staff and 26 people from Samu between 9 and 12 months after the events.

Based on the expertise of Public Health France and the model developed for the ESPA study on November 13th, the Public Health Department of the University Hospital of Nice wished to carry out a specific study among the health professionals of the University Hospital of Nice and the Hospitals pediatrics of Nice CHU-Lenval, as well as students of the Faculty of Medicine of Nice Sophia-Antipolis.

Many professionals of all categories were directly impacted: either at the scene of the attack as a civilian population or as professionals, or in the care services that received the victims and families (including services of the Pasteur2 hospital, Lenval Hospital on the Promenade des Anglais).

The population of medical students is also included in the study, and external students in particular have made a significant contribution to the Institut Médico-Légal.

This involvement could be done directly (presence as hospital staff at the scene of the attack, care of the victims or their relatives, in the emergency and care services), but also indirect (close and knowledge affected by the attack, specific repercussions in the local context, forced changes in the organization of work). It is therefore all hospital professionals, medical students (external, internal) and paramedical students who will be involved in the study.

ELIGIBILITY:
* inclusion criteria: hospital staff Whether or not directly involved in the attack of 14 July 2016.
* exclusion criteria: non hospital staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The staff
  * From the establishments of the Nice University Hospital: Hôpital Pasteur, Hôpital l' Archet, Hôpital de Cimiez, Hôpital St Roch, Unité centrale de production or UCP, Hôpital de Tende.
  * From the Lenval Hospital building: staff of the Nice CHU-Lenval Children's Hospital, and staff of the Lenval Foundation.
  * Students (external from M1 onwards, i. e. the 4th year, and interns) enrolled in Nice-Sophia Antipolis Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
questionnaire about health impact | 1 year
  document the health impact of these events and provide useful information for the care arrangements for the populations involved and in the event of a new attack.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No